CLINICAL TRIAL: NCT04834297
Title: Prapela™ SVS: A Cost-effective Stochastic Vibro-tactile Stimulation Device to Improve the Clinical Course of Infants With Neonatal Opioid Withdrawal Syndrome.
Brief Title: Use of SVS Device to Improve Outcomes for Neonatal Opioid Withdrawal Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001552
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Opioid Withdrawal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SVS mattress (Experimental): Infants randomized to the experimental arm will have the SVS mattress placed in their crib within 48 hours of birth and will continue till discharge home after the completion of monitoring phase of NOWS or till determination is made to initiate pharmacotherapy for NOWS.
  Interventions: Other: Prapela SVS mattress
- Standard mattress (No Intervention): Infants randomized to the no intervention arm will continue to be cared for using the standard hospital crib mattress throughout their birth hospitalization.

INTERVENTIONS:
Other: Prapela SVS mattress — The intervention will be using the Prapela SVS crib mattress to complement non-pharmacological management of NOWS for the purposes of prevention of pharmacological treatment of NOWS
  Arms: SVS mattress

SUMMARY:
Maternal use and addiction to opioids has resulted in an unprecedented rise in drug withdrawal complications in newborns known as neonatal opioid withdrawal syndrome (NOWS), also referred to as neonatal abstinence syndrome (NAS). Between 2004 and 2016, NOWS admissions increased more than fourfold with an average hospital stay nearly 3.2 times longer (15.9 hospital days compared with 4.98) than for a non-NOWS patient resulting in a surge in annual costs to almost $573 million with 83% attributed to state Medicaid programs. While there is no accepted standard for treating NAS, non-pharmacological bundles are recommended, as an initial course of treatment moving to pharmacological care when required. Unfortunately, non-pharmacological care (swaddling, rocking, frequent feedings, and skin contact) require significant use of human resources. To reduce the increasing burden on limited resources, the evidence emerges that hospitals are trying to adapt baby products for consumers that were neither intended nor tested for use in NAS infants as part of their non-pharmacological bundle. The objective of this application is to establish the safety, efficacy, and acceptability of our hospital bassinet pad with stochastic vibrotactile stimulation (SVS) technology as an adjunctive, non-pharmacological treatment to improve the care of infants with NOWS. To accomplish the objective, the investigators plan to execute the following specific aims; 1) determine the efficacy of the SVS hospital bassinet pad, 2) demonstrate the safety of the SVS hospital bassinet pad, and 3) assess acceptability of the device with clinical staff and parents caring for infants with NOWS. The successful completion of the project will provide data to support FDA clearance for commercialization of this low-cost, non-pharmacological device to improve the clinical course of newborns with NOWS.

DETAILED DESCRIPTION:
In preliminary work using a research grade device, the investigators tested stochastic vibrotactile stimulation (SVS) in infants with NOWS. Twenty six full term infants who were opioid exposed, as determined by meconium drug screening tests and/or maternal self-report, were studied. Infants were excluded if any of the following characteristics were present: congenital abnormality, anatomic brain abnormality, hydrocephalus, intraventricular hemorrhage > grade 2, seizure disorder not related to withdrawal, significant cardiac shunt, anemia and/or infection. Using a single session, within-subject design characteristics were compared during periods on and off SVS. Movement, heart rate, respiratory rate, temperature and oxygen saturation were quantified by continuous physiologic measurement. Infants were between 38.3 and 44.7 weeks at the time of study. This novel work demonstrated that SVS reduced prolonged movement activity and improved cardiorespiratory function in the opioid-exposed neonates with 35% reduction in movement and significant reductions in tachypnea and tachycardia. There were no noted adverse effects; specifically no alterations in temperature control or oxygen saturation. Parents and nurses reported that infants seemed less irritable, calmer, and slept better.

Specific Aim #1: To determine the efficacy of the Prapela SVS device in preventing the need for pharmacologic treatment in term infants ≥35 weeks gestation with prenatal opioid exposure.

Hypotheses:

1A. The use of the Prapela SVS device will reduce the need for pharmacologic treatment for NOWS by 22.5%.

1B. The Prapela SVS device will reduce periods of cries characterized as fussy and pain in the two study groups.

1.1 1A. Study Intervention and Timing: Parents of infants at risk for NOWS will be approached for consent within the first 48 hours after birth prior to manifestation of withdrawal symptoms. After informed written consent is obtained the study procedures will be initiated. SVS will be delivered with a specially-constructed mattress developed during Phase I of the SBIR that delivers gentle, random, low-level stimulation (30-60 Hz, 10-12 micrometers RMS) in continuously. SVS will be added to existing non-pharmacologic care within the first 24 hours of birth until day 5 or until pharmacologic treatment is initiated. The rationale for the selection of this experimental window are: 1. Majority of infants do not start manifesting signs of NOWS prior to 48hours of life. 2. Most infants who require treatment with opioids for severe withdrawal typically begin treatment on day 3 to 5 of life. 3. To test the efficacy of the SVS device, we seek to study the infant who has not yet manifested signs of NOWS and determine if it is safe and effective in preventing the need for pharmacotherapy. All infants enrolled will remain on the SVS mattress throughout the first 5 days of life or until pharmacologic treatment is started except for periods of care and feeding. The use of infant swings or other motion devices will be prohibited once enrolled in the study. Two thirds (80 infants) will be randomized to receive the SVS mattress and one-third (40 infants) will receive standard care only.

1. B Maternal and infant clinical characteristics: Clinical characteristics of the mother and infant will be abstracted from the medical record by a trained research coordinator using standardized definitions. Modified Finnegan scores or Eat, Sleep and Console (ESC) score will be abstracted from the medical record and summed over each 24 hour period. The nursing team providing clinical care to these infants are trained in using both the scoring tools. Caregiver's assessment of infant state will be recorded every 6 hours in a bedside diary. Missing data will be explicitly noted.

1C. Environmental and physiological measurements: Analyses of Cry Characteristics: To further characterize the ability of the SVS device to soothe infants with NOWS, we will utilize novel technology developed and patented by Dr. Ariana Anderson at UCLA called the ChatterBaby. Her work is based on the known association of abnormal cry with abnormal central nervous system development or disease. A more recent version of the ChatterBaby cry detection and cry translation algorithms will be used for this study. These algorithms are trained against hours of non-cry data, including NICU ambient sound, to robustly identify crying periods by automation. The cry during three primary states (fussy, hungry, pain) will be quantified and analyzed between the two groups.

Specific Aim #2: Demonstrate the safety of the SVS hospital bassinet for infants with NOWS.

2. Hypothesis: The device will meet non-clinical safety standards required for FDA clearance.

Additionally, non-clinical studies (including electrical, thermal safety, biocompatibility, and electromagnetic compatibility) will be completed to verify the device meets or exceeds safety requirements for FDA clearance. Sampling before and after clinical use, as well as durability testing will be performed to ensure that the devices deliver the specified vibration over time. Prapela has prepared a data development plan (DDP) that aligns with the proposed measures to mitigate the identified risks to health of the Prapela® SVS Hospital Bassinet Pad.

Specific Aim #3: Assess the acceptability of the SVS mattress to infants' mothers and nurses.

Hypothesis: The Prapela SVS device will be accepted and valued by both nursing caregivers and parents.

A questionnaire will be administered at the end of the experimental period to both the nursing staff present on the final shift of the period and to the mother, or other care-giver if mother not able to be present.

ELIGIBILITY:
Inclusion Criteria:

1. Infants ≥ 35 weeks gestation with prenatal opioid exposure

Exclusion Criteria:

1. Infants < 35 weeks gestational age at birth
2. Infants receiving opioids for non-NOWS indications
3. Infants with congenital anomalies
4. Infants with known central nervous system anomalies
5. Infants with seizures unrelated to opioid withdrawal
6. Infants with hydrocephalus
7. Infants with intraventricular hemorrhage ≥ grade 2 (Papille Scale)
8. Infants with severe anemia (hemoglobin < 8)
9. Infants with suspected and/or confirmed infection
10. Infants deemed to be clinically unstable by their medical provider
11. Multiple births

Ages: 0 Days to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Number of participants requiring pharmacologic treatment of NOWS | Baseline up to Day 5 of life
  All the infants enrolled in the study will be assessed for the need of pharmacological management of NOWS with initiation of morphine sulfate, based on either the modified Finnegan score or ESC tool.

SECONDARY OUTCOMES:
Mean daily percentage of time characterized as pain or fussy crying | Baseline up to day 5 of life
  This outcome is calculated as the total daily duration of crying categorized as pain or fussy by the ChatterBaby algorithm, divided by 24 hours. For each participant, we will consider the daily percentage of time characterized as pain or fussy crying, from randomization to Day 5 of life or initiation of pharmacologic treatment for NOWS (whichever occurs first). This will be analyzed using mixed effects linear regression models.
Mean modified Finnegan score | Baseline up to day 5 of life
  The modified Finnegan score is measured on a scale from 0 to 45. Larger scores indicate more severe symptoms of withdrawal. For participants assessed with the modified Finnegan score, we will consider the daily average score, from randomization to Day 5 of life or initiation of pharmacologic treatment for NOWS. We will analyze the repeated measures of the daily average modified Finnegan score by using mixed effects linear regression models.
Mean ESC score | Baseline up to day 5 of life
  An ESC score will be calculated based on the count of symptoms present on the assessment tool, ranging from 0 to 3. Larger scores indicate more severe symptoms of withdrawal. For participants assessed with the ESC tool, we will consider the daily average score, from randomization to Day 5 of life or initiation of pharmacologic treatment for NOWS. We will analyze the repeated measures of the daily average ESC score by using mixed effects linear regression models.
Mean number of days until readiness for hospital discharge | Duration of hospital stay, an expected average of 11 days
  Measured as the number of days to readiness of discharge from hospital. We will compare the distributions of the number of days until readiness for discharge by using a negative binomial regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Rachana Singh, MD, MS, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh R, Trinquart L, Koethe B, Cordova M, Rhein L, Bibi S, Fey J, Anderson A, Davis JM. Efficacy of stochastic vibro-tactile stimulation for newborns at risk of neonatal opioid withdrawal syndrome. Pediatr Res. 2025 May 23. doi: 10.1038/s41390-025-04162-2. Online ahead of print. PMID 40410582